CLINICAL TRIAL: NCT02070484
Title: Efficacy of a Human Amniotic Tissue-derived Allograft, NuCel, in Patients Undergoing Posteriolateral Lumbar Fusions for Degenerative Disc Disease
Brief Title: Human Amniotic Tissue-derived Allograft, NuCel, in Posteriolateral Lumbar Fusions for Degenerative Disc Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: OhioHealth (Other)
Collaborators: NuTech Medical, Inc (Industry)
Responsible Party: Principal Investigator, Joseph A. Shehadi, MD, Principal Investigator, OhioHealth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OH2-13-0034
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Lumbar Degenerative Disc Disease; Spinal Stenosis; Spondylolisthesis; Spondylosis; Intervertebral Disk Displacement; Intervertebral Disk Degeneration; Spinal Diseases; Bone Diseases; Musculoskeletal Diseases; Spondylolysis
Keywords: NuCel; Lumbar Spine; Degenerative Disease; Efficacy; Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis; Spondylolisthesis; Spondylosis; Intervertebral Disc Displacement; Spinal Diseases; Bone Diseases; Musculoskeletal Diseases; Spondylolysis | interventions — Grafton demineralized bone matrix gel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NuCel (Experimental): Stemcell allograft
  Interventions: Biological: NuCel
- Demineralized Bone Matrix (DBM) (Active Comparator): Demineralized Bone Matrix (DBM) bone graft substitute
  Interventions: Biological: Demineralized Bone Matrix

INTERVENTIONS:
Biological: NuCel
  Arms: NuCel
Biological: Demineralized Bone Matrix
  Arms: Demineralized Bone Matrix (DBM)

SUMMARY:
The purpose of this study is to compare the effect and safety of NuCel to DBX on patients undergoing posteriolateral lumbar spinal fusions for degenerative disc disease.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 75 years
* Symptomatic, single-level degenerative lumbar disc disease, spondylosis or spondylolisthesis
* Failed conservative treatments
* Low risk for non-union
* Must be candidates for single-level, posteriolateral lumbar spine fusion
* Must be able and willing to give Informed Consent
* English-speaking

Exclusion Criteria:

* Smoker (any smoking ≤3 months prior to consent); (Patel et al. 2013)
* Patients with poorly controlled diabetes mellitus (HgbA1c > 7%)
* Documented osteoporosis
* Prior lumbar spinal surgery at the same spinal level, or immediately adjacent spine level, to the level being operated on
* Back pain due to infection, tumour, or metabolic bone disease
* Terminal disease, such as HIV infection, neoplasm
* Autoimmune disease, such as rheumatoid arthritis
* Morbid obesity (body mass index (BMI) of 35 kg/m2)
* Major psychiatric illness in the last year
* History of alcohol or drug abuse in the last year
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02; Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Shehadi, MD, Principal Investigator — OhioHealth
Locations (2):
- United States (2):
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- NuCel: Stemcell allograft
  NuCel
- Demineralized Bone Matrix (DBM): Demineralized Bone Matrix (DBM) bone graft substitute
  Demineralized Bone Matrix
Period: Overall Study
Arm/Group | NuCel | Demineralized Bone Matrix (DBM)
Started | 3 | 3
Completed | 2 | 3
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NuCel | Demineralized Bone Matrix (DBM) | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Oswestry Disability Index [Mean (Full Range); unit: units on a scale] — The Oswestry Disability Index (ODI) measures disability on a scale of 0-100, where higher scores correspond to greater disability.
  units on a scale | 28.7 [26 to 32] | 26.7 [19 to 34] | 27.7 [19 to 34]

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Disability Index
Description: The Oswestry Disability Index (ODI) measures disability on a scale of 0-100, where higher scores correspond to greater disability.
Time Frame: 12 months
Population: One of three NuCel patients withdrew before 12 months; therefore, analysis comprises two NuCel patients and three DBM patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NuCel | Demineralized Bone Matrix (DBM)
Number analyzed (Participants) | 2 | 3
units on a scale | 8.0 (11.3) | 15.3 (17.2)

2. Secondary Outcome: Computed Tomography (CT) Scans to Assess Lumbar Bone Fusion
Description: CT scans reviewed by an independent radiologist and scored according to three categories: no fusion, any fusion, solid fusion.
Time Frame: 6 and 12 months
Population: The study was terminated due to low enrollment; therefore, CT scans at 6 and 12 months were not conducted.
Arm/Group | NuCel | Demineralized Bone Matrix (DBM)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Oswestry Disability Index
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NuCel | Demineralized Bone Matrix (DBM)
Number analyzed (Participants) | 3 | 3
units on a scale | 28.7 (3.1) | 26.7 (7.5)

4. Primary Outcome: Oswestry Disability Index
Description: as for outcome 1
Time Frame: 1 month
Population: One of three NuCel patients withdrew; therefore, analysis comprises two NuCel patients and three DBM patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NuCel | Demineralized Bone Matrix (DBM)
Number analyzed (Participants) | 2 | 3
units on a scale | 15.5 (12.0) | 26.7 (13.7)

5. Primary Outcome: Oswestry Disability Index
Description: as for outcome 1
Time Frame: 2 months
Population: One of three NuCel patients withdrew; therefore, analysis comprises two NuCel patients and three DBM patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NuCel | Demineralized Bone Matrix (DBM)
Number analyzed (Participants) | 2 | 3
units on a scale | 19.5 (17.7) | 22.0 (9.6)

6. Primary Outcome: Oswestry Disability Index
Description: as for outcome 1
Time Frame: 3 months
Population: One of three NuCel patients withdrew; therefore, analysis comprises two NuCel patients and three DBM patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NuCel | Demineralized Bone Matrix (DBM)
Number analyzed (Participants) | 2 | 3
units on a scale | 10.0 (12.7) | 25.7 (7.5)

7. Primary Outcome: Oswestry Disability Index
Description: as for outcome 1
Time Frame: 6 months
Population: One of three NuCel patients withdrew; therefore, analysis comprises two NuCel patients and three DBM patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NuCel | Demineralized Bone Matrix (DBM)
Number analyzed (Participants) | 2 | 3
units on a scale | 7.5 (9.2) | 14.7 (10.6)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded through 12 months post-operatively
Arm/Group | NuCel | Demineralized Bone Matrix (DBM)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NuCel (N=3) | Demineralized Bone Matrix (DBM) (N=3)
Prolonged hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) — Intermittent diarrhea, bloating, and stomach pain beginning post-operative day 5. Symptoms improved with bowel regimen and liquid diet; solid food resumed post-operative day 5. Patient discharged post-operative day 5.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT02070484/Prot_SAP_000.pdf